CLINICAL TRIAL: NCT01029171
Title: "Action Seniors!: A 12 Month Randomized Controlled Trial of a Home Based Strength and Balance Retraining Program in Reducing Falls.
Brief Title: Action Seniors! Exercise to Prevent Falls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Teresa Liu-Ambrose, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H04-70171
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Falls
Keywords: falls; balance training; strength training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): OEP (Otago Exercise Program; home-based balance and strength retraining program)
  Interventions: Behavioral: Home-based balance and strength retraining exercise program.
- 2 (Active Comparator): CON (control; usual care)
  Interventions: Behavioral: control; usual care

INTERVENTIONS:
Behavioral: Home-based balance and strength retraining exercise program. — A 12-month home-based balance and strength restraining program delivered by a physical therapist
  Arms: 1
Behavioral: control; usual care — Usual care as prescribed by geriatrician.
  Arms: 2

SUMMARY:
This study will be a randomized controlled trial to determine the efficacy of the Otago Exercise Program (OEP) on falls among seniors with a history of falls.

DETAILED DESCRIPTION:
A total of 344 community-dwelling adults aged 70 years and older who are referred to a falls clinic secondary to seeking medical attention due to a fall will be randomized to either the 12-month OEP group or usual care. There will be three measurement sessions: baseline, 6 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Adults older than or 70 years attending a Falls Prevention Clinic Service;
2. Understands, speaks, and reads English proficiently;
3. MMSE 8 score > 24/30;
4. Had one documented non-syncopal fall in the last 12 months and one of the following: a) A Physiological Profile Assessment (PPA) score of at least 1 SD above normal; OR 2) Timed Up and Go Test (TUG) performance of greater than 15 seconds; OR 3) One additional documented non-syncopal fall in the previous 12 months;
5. Expected to live greater than 12 months;
6. Community-dwelling (i.e., not residing in a nursing home, extended care unit, or assisted-care facility);
7. Able to walk 3 meters with or without an assistive device; and
8. Able to provide written informed consent.

Exclusion Criteria:

1. Diagnosed with a neurodegenerative disease (e.g., Parkinson's disease);
2. Diagnosed with dementia (of any type);
3. Had a stroke;
4. Have clinically significant peripheral neuropathy or severe musculoskeletal or joint disease; or
5. Have a history indicative of carotid sinus sensitivity (i.e., syncopal falls).

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 344 (Actual)
Dates: Start 2009-11; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Falls over a 12 month period. | 12 months

SECONDARY OUTCOMES:
Secondary outcomes of interest include: 1) physiological falls risk; 2) mobility; 3) cognitive function; and 4) economic evaluation. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Liu-Ambrose, Principal Investigator — University of British Columbia; Karim Khan, Ph.D, Study Director — University of British Columbia; Larry Dian, MD, Study Director — University of British Columbia; Wendy Cook, MD, Study Director — University of British Columbia; Penny Brasher, Ph.D, Study Director — University of British Columbia; Carlo Marra, Ph.D, Study Director — University of British Columbia; Jennifer Davis, Ph.D, Study Director — University of British Columbia
Locations (1):
- Aging, Mobility, and Cognitive Neuroscience Laboratory, Vancouver Falls Prevention Clinic, University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Falck RS, Hsu CL, Davis JC, Rice J, Dao E, Dian L, Madden K, Skelton DA, Parmar N, Cook WL, Khan KM, Liu-Ambrose T. Effect of a home-based exercise program on subsequent falls among community-dwelling older adults with cognitive frailty: A sub-group analysis of a randomized controlled trial. Maturitas. 2025 Jan;191:108151. doi: 10.1016/j.maturitas.2024.108151. Epub 2024 Nov 7. PMID 39561465
- [Derived] Davis JC, Hsu CL, Ghag C, Starkey SY, Jacova P, Dian L, Parmar N, Madden K, Liu-Ambrose T. Baseline health-related quality of life predicts falls: a secondary analysis of a randomized controlled trial. Qual Life Res. 2022 Nov;31(11):3211-3220. doi: 10.1007/s11136-022-03175-2. Epub 2022 Jul 7. PMID 35798988
- [Derived] Davis JC, Hsu CL, Barha C, Jehu DA, Chan P, Ghag C, Jacova P, Adjetey C, Dian L, Parmar N, Madden K, Liu-Ambrose T. Comparing the cost-effectiveness of the Otago Exercise Programme among older women and men: A secondary analysis of a randomized controlled trial. PLoS One. 2022 Apr 20;17(4):e0267247. doi: 10.1371/journal.pone.0267247. eCollection 2022. PMID 35442974
- [Derived] Liu-Ambrose T, Davis JC, Falck RS, Best JR, Dao E, Vesely K, Ghag C, Rosano C, Hsu CL, Dian L, Cook W, Madden KM, Khan KM. Exercise, Processing Speed, and Subsequent Falls: A Secondary Analysis of a 12-Month Randomized Controlled Trial. J Gerontol A Biol Sci Med Sci. 2021 Mar 31;76(4):675-682. doi: 10.1093/gerona/glaa239. PMID 33225343
- [Derived] Davis JC, Khan KM, Hsu CL, Chan P, Cook WL, Dian L, Liu-Ambrose T. Action Seniors! Cost-Effectiveness Analysis of a Secondary Falls Prevention Strategy Among Community-Dwelling Older Fallers. J Am Geriatr Soc. 2020 Sep;68(9):1988-1997. doi: 10.1111/jgs.16476. Epub 2020 May 29. PMID 32472567
- [Derived] Liu-Ambrose T, Davis JC, Best JR, Dian L, Madden K, Cook W, Hsu CL, Khan KM. Effect of a Home-Based Exercise Program on Subsequent Falls Among Community-Dwelling High-Risk Older Adults After a Fall: A Randomized Clinical Trial. JAMA. 2019 Jun 4;321(21):2092-2100. doi: 10.1001/jama.2019.5795. PMID 31162569
- [Derived] Liu-Ambrose T, Davis JC, Hsu CL, Gomez C, Vertes K, Marra C, Brasher PM, Dao E, Khan KM, Cook W, Donaldson MG, Rhodes R, Dian L. Action seniors! - secondary falls prevention in community-dwelling senior fallers: study protocol for a randomized controlled trial. Trials. 2015 Apr 10;16:144. doi: 10.1186/s13063-015-0648-7. PMID 25873254